CLINICAL TRIAL: NCT06720207
Title: Exploratory Study on the Efficacy of 68Ga-Pentixafor PET/MR in Detecting Lesions in Non-Hodgkin Lymphoma and Multiple Myeloma
Brief Title: Efficacy of 68Ga-Pentixafor PET/MR in Detecting Non-Hodgkin Lymphoma and Multiple Myeloma Lesions
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SEH-2024210
Record Dates: First submitted 2024-11-27; First posted 2024-12-06 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2024-12

CONDITIONS: Non Hodgkin's Lymphoma; Multiple Myeloma (MM)
Keywords: PET/MR; Non Hodgkin's Lymphoma; multiple myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Research group: It is expected to include 30 newly diagnosed NHL or MM patients, and the tracer radiation used in the study is extremely small and will not have any physiological effects on the subjects.

SUMMARY:
In this study, the investigators intend to utilize 68Ga-Pentixafor Positron Emission Tomography（PET） imaging for patients diagnosed with non-Hodgkin lymphoma (NHL) and multiple myeloma (MM). The investigators will compare the imaging results with those obtained from 18F-FDG imaging, and a correlation analysis will be performed to assess progression-free survival among patients. This analysis aims to evaluate the diagnostic efficacy and the potential for early prediction of treatment efficacy associated with 68Ga-Pentixafor in these specific conditions.

DETAILED DESCRIPTION:
The hematolymphatic system comprises blood, lymph nodes, extranodal lymphatic tissues, bone marrow, and the spleen. When malignant transformations occur within this system, they often infiltrate various tissues and organs throughout the body. Therefore, a comprehensive assessment of all tissues and organs is necessary to delineate the lesions' extent and conduct clinical staging to guide treatment. Lymphoma is the most prevalent malignancy of the hematologic system, with non-Hodgkin lymphoma (NHL) accounting for a significant incidence within this category, representing approximately 90% of lymphomas in our country. The clinical classification of NHL is complex, exhibiting considerable heterogeneity in biological behavior, immunophenotyping, and prognosis. The main subtypes include diffuse large B-cell lymphoma (DLBCL), follicular lymphoma (FL), T-cell lymphoma (TCL), marginal zone lymphomas (MZL), and mantle cell lymphoma (MCL). Multiple myeloma (MM) is a malignant disease characterized by the clonal proliferation of abnormal plasma cells and is the second most common hematologic malignancy following lymphoma. Common symptoms include organ dysfunction related to myeloma, encapsulated in the "CRAB" criteria-hypercalcemia, renal insufficiency, anemia, and bone disease-along with manifestations of organ damage due to amyloidosis. The prognosis is poor if patients do not receive timely and effective treatment.

Chemokine receptor 4 (CXCR4) is a member of the C-X-C motif (CXC) subfamily of chemokine receptors and is widely expressed in various types of organ tissue. It significantly regulates numerous physiological processes through interaction with CXC-chemokine ligand 12 (CXCL12). The CXCR4/CXCL12 biological axis is critical in the proliferation, invasion, and metastasis of NHL and MM and is considered a marker of poor prognosis. Recently, a new positron emission tomography (PET) tracer targeting CXCR4, 68Ga-Pentixafor, has been developed and is being increasingly utilized to diagnose hematological malignancies. The 68Ga-Pentixafor PET demonstrates notable advantages in identifying lymphoma, particularly indolent types, as well as in detecting early small lesions associated with MM. It shows greater sensitivity compared to 18F-fluorodeoxyglucose (FDG) imaging. This advancement not only enhances patient diagnosis and efficacy evaluation but also functions as a biological targeting molecule for individuals with poor prognostic outcomes, enabling these patients to access more intensive treatment options.

18F-fluorodeoxyglucose (FDG) is the most widely used tracer in nuclear medicine for tumor imaging, applicable to the initial staging and efficacy assessment of the vast majority of tumors. According to the 2021 guidelines from the Chinese Medical Association's Nuclear Medicine Branch and recommendations from the International Myeloma Working Group (IMWG), 18F-FDG positron emission tomography / computed tomography (PET/CT) imaging is recommended for the diagnostic and therapeutic management of all lymphoma and MM patients. However, it is important to note that the uptake of FDG in NHL is related to its pathological type; DLBCL and FL typically exhibit high FDG uptake, while MZL, MCL, and small lymphocytic lymphoma(SLL) usually show moderate to low FDG uptake. This variability results in differences in the diagnostic accuracy of 18F-FDG PET depending on the subtype of NHL. Additionally, approximately 11% of MM patients may present with false-negative FDG imaging, which could be attributed to factors such as small lesion size, a lower proliferation rate of clonal plasma cells, or hexokinase deficiency. Furthermore, physiological or inflammatory uptake of 18F-FDG can sometimes interfere with the detection of MM lesions.

In summary, early diagnosis before treatment, precise staging, and post-treatment prognostic stratification, as well as the detection of residual tumor metabolic activity, represent significant challenges in the diagnosis and treatment of NHL and MM. The use of 68Ga-pentixafor PET/MR allows for non-invasive visualization of CXCR4 expression in vivo, demonstrating high sensitivity for NHL and MM with low FDG uptake. This capability enhances diagnostic accuracy and facilitates precise staging, contributing to the development of personalized treatment plans and ultimately improving patient outcomes. Through the implementation of this project, the investigators aim to introduce new technologies in the management of NHL and MM patients, providing more effective diagnostic and therapeutic options.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 years or older
2. ECOG < 2
3. Newly diagnosed patients with NHL and MM who have been confirmed or are highly suspected based on pathological examination
4. Completion of 18F-FDG PET/CT or PET/MR imaging within the past week in our department

Exclusion Criteria:

1. Pregnant and breastfeeding women;
2. Individuals with severe hepatic and renal failure;
3. Patients with concurrent malignancies;
4. Individuals unable to remain supine for a duration of 30 minutes to complete the examination;
5. Patients with diagnosed claustrophobia;
6. Patients containing metallic implants;
7. Individuals deemed unsuitable for participation in clinical trials by researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who meet the inclusion and exclusion criteria and are willing to follow the research process.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Ann Arbor staging | After the patient signs the informed consent form and completes the scan, an average of 2 days.
  All patients were classified into stages I-IV based on Ann Arbor staging according to visual methods.
Metabolic parameters | After the patient signs the informed consent form and completes the scan, an average of 2 days.
  Calculate maximum standardized uptake value (SUVmax (lesion)) of all affected lymphoma and extranodal organs. Set a region of interest with a diameter of approximately 10mm in the descending segment of the thoracic aorta, calculate the standardized uptake value (SUVmean) of the mediastinal blood pool, calculate SUVmax (lesion)/SUVmean (blood pool).

IPD SHARING:
Plan to Share IPD: No
For the protection of patient privacy, we will not share patient information, but other researchers can apply through the project contact person if they have reasonable reasons.